CLINICAL TRIAL: NCT00093197
Title: Intracoronary KAI-9803 for Injection as an Adjunct to Primary Percutaneous Coronary Intervention for Acute ST-Elevation Myocardial Infarction
Brief Title: Safety of KAI-9803 for Injection With Angioplasty Following Heart Attack
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: KAI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KAI-9803-001
Record Dates: First submitted 2004-10-04; First posted 2004-10-07 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-08

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — KAI 9803; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A1: KAI-9803 (Experimental)
  Interventions: Drug: KAI-9803 for Injection
- A2: KAI-9803 (Experimental)
  Interventions: Drug: KAI-9803 for Injection
- A3: KAI-9803 (Experimental)
  Interventions: Drug: KAI-9803 for Injection
- A4: KAI-9803 (Experimental)
  Interventions: Drug: KAI-9803 for Injection
- A5: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KAI-9803 for Injection — 0.05 mg
  Arms: A1: KAI-9803
Drug: KAI-9803 for Injection — 0.5 mg
  Arms: A2: KAI-9803
Drug: KAI-9803 for Injection — 1.25 mg
  Arms: A3: KAI-9803
Drug: KAI-9803 for Injection — 5 mg
  Arms: A4: KAI-9803
Drug: Placebo
  Arms: A5: Placebo

SUMMARY:
Restoring blood flow to coronary arteries as quickly as possible is the best way to reduce the damage to the muscle that occurs with a heart attack. However, up to 25-50% of patients who have angioplasty may have ongoing damage to the heart muscle when the blockage is opened and blood flow is restored. Complications which may result from this ongoing damage include a larger area of damaged muscle in the heart, enlargement of the heart, an increased risk of death, and an increased risk of heart failure. Some of the ongoing damage may involve increased levels of the protein kinase C (PKC) enzyme. KAI-9803 is a selective inhibitor of delta PKC. In this study, delta PKC is used with angioplasty and other standard procedures to restore blood flow after a heart attack. This study is designed to evaluate safety of different amounts of KAI-9803 when used in treating heart attack patients undergoing angioplasty. We will also try to evaluate whether KAI-9803 can reduce the amount of heart muscle damage and the complications that may occur in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of cardiac ischemia at rest or with increasing frequency (angina or angina equivalent), with episodes lasting for at least 30 minutes within 6 hours of presentation
* Persistent ST-segment elevation of ≥ 0.2 mV in at least 2 contiguous precordial leads indicative of anterior Myocardial Infarction (MI) location (leads V1-V4)
* At least 18 years old
* Complete occlusion of the left anterior descending artery (Thrombolysis in Myocardial Infarction (TIMI) 0-1 flow) demonstrated on the initial angiogram
* Culprit lesion suitable for primary percutaneous coronary intervention (PCI)

Exclusion Criteria:

* Any left bundle branch block (new or old), intraventricular conduction defect, or paced rhythm that would obscure the diagnosis of acute anterior ST Elevation Myocardial Infarction (STEMI)
* Any prior documented myocardial infarction (MI), including old Q waves documented on prior ECGs or a clinical history of definite MI
* Any prior coronary artery bypass grafting (CABG)
* Cardiogenic shock at initial hospital presentation, consisting of persistent hypotension (systolic blood pressure < 90 mm Hg for > 20 minutes) and signs of end-organ dysfunction (oliguria, altered mental status, poor peripheral perfusion, and lactic acidosis)
* TIMI grade 2 or 3 flow in the left anterior descending artery documented on the initial diagnostic angiogram
* Culprit lesion in the left anterior descending artery that is not suitable for primary PCI
* Treatment with intravenous fibrinolytic therapy (i.e. alteplase, reteplase, tenecteplase, or streptokinase) within the 24 hours before presentation
* Pregnancy
* Know baseline creatinine > 2.5 mg/dL without renal dialysis/renal replacement therapy within the 30 days before presentation
* Inability to comply with study procedures, inability to undergo cardiac catheterization or primary percutaneous coronary intervention (PCI)
* Participation in a study of experimental therapy (drug or device) within 30 days of presentation, or prior participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2004-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 30 days
Number of participants with major cardiac events (death, congestive heart failure, recurrent myocardial infarction, repeat target vessel revascularization) | 6 months

SECONDARY OUTCOMES:
Creatine kinase-myocardial band (CK-MB) | 7 days or hospitalization discharge, whichever occurs first
ST-segment elevation | 24 hours
Angiography vessel flow | Day 1
Infarct size by single photon emission computed tomography (SPECT) | 14 days
Echocardiographic left ventricular ejection fraction (LVEF) | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Clinical Research Institute, Durham, North Carolina, United States